CLINICAL TRIAL: NCT02746991
Title: A Multi-center, Controlled, Safety and Efficacy Study of a Fluocinolone Acetonide Intravitreal (FAI) Insert in Subjects With Chronic Non-infectious Uveitis Affecting the Posterior Segment of the Eye
Brief Title: Safety and Efficacy Study of a FAI Insert in Subjects With Chronic Non-infectious Posterior Uveitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSV-FAI-005
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Posterior Uveitis; Intermediate Uveitis; Panuveitis
MeSH Terms: conditions — Uveitis, Posterior; Uveitis, Intermediate; Panuveitis | interventions — salicylhydroxamic acid; Fluocinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Injection (Sham Comparator): Sham Injection
  Interventions: Drug: Sham Injection
- FAI Insert (Experimental): FAI Insert (0.18 mg fluocinolone acetonide)
  Interventions: Drug: FAI Insert

INTERVENTIONS:
Drug: Sham Injection — Placebo
  Other Names: Placebo
  Arms: Sham Injection
Drug: FAI Insert — Fluocinolone Acetonide
  Other Names: Fluocinolone Acetonide
  Arms: FAI Insert

SUMMARY:
Phase 3, multi-center, randomized, masked, controlled study to evaluate the safety and efficacy of an injectable fluocinolone acetonide intravitreal (FAI) insert for the management of subjects with chronic non-infectious uveitis affecting the posterior segment of the eye. Patients will be randomized to receive either a sham injection or the FAI insert and will be observed for three years following treatment.

DETAILED DESCRIPTION:
This is a phase 3, multi-center, randomized, masked, controlled study to evaluate the safety and efficacy of an injectable fluocinolone acetonide intravitreal (FAI) insert for the management of subjects with chronic non-infectious uveitis affecting the posterior segment of the eye. Patients will be randomized to receive either a sham injection or the FAI insert and will be observed for three years following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or non pregnant female at least 18 years of age at time of consent
* One or both eyes having a history of recurrent non-infectious uveitis affecting the posterior segment of the eye with or without anterior uveitis > 1 year duration
* At the time of enrollment (Day 1), study eye has < 10 anterior chamber cells/High Power Field (HPF) and a vitreous haze ≤ grade 2.
* Visual acuity of study eye is at least 15 letters on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart
* Subject is not planning to undergo elective ocular surgery during the study
* Subject has ability to understand and sign the Informed Consent Form
* Subject is willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
* During the 12 months prior to enrollment (Day 1), the study eye has either received treatment:

  * systemic corticosteroid or other systemic therapies given for at least 3 months, and/or
  * at least 2 intra- or peri-ocular administrations of corticosteroid for management of uveitis

OR the study eye has experienced recurrence:

• at least 2 separate recurrences of uveitis requiring systemic, intra- or peri-ocular injection of corticosteroid

Exclusion Criteria:

* Allergy to fluocinolone acetonide or any component of the Fluocinolone Acetonide Intravitreal (FAI) insert
* History of posterior uveitis only that is not accompanied by vitritis or macular edema
* History of iritis only and no vitreous cells, anterior chamber cells or vitreous haze
* Uveitis with infectious etiology
* Vitreous hemorrhage
* Intraocular inflammation associated with a condition other than noninfectious uveitis (e.g. intraocular lymphoma)
* Ocular malignancy in either eye, including choroidal melanoma
* Toxoplasmosis scar in study eye or scar related to previous viral retinitis
* Previous viral retinitis
* Current viral diseases of the cornea and conjunctiva including epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, and varicella, mycobacterial infections of the eye or fungal diseases of ocular structures
* Media opacity precluding evaluation of retina and vitreous
* Peripheral retinal detachment in area of insertion
* Diagnosis of any form of glaucoma or ocular hypertension in study eye at Screening, unless study eye has been previously treated with an incisional surgery procedure that has resulted in stable Intraocular pressure (IOP) in the normal range (10-21 mmHg)
* IOP > 21 mmHg or concurrent therapy at Screening with any IOP-lowering pharmacologic agent in the study eye
* Chronic hypotony (< 6 mmHg)
* Ocular surgery on the study eye within 3 months prior to study Day 1
* Capsulotomy in study eye within 30 days prior to study Day 1
* Prior intravitreal treatment of study eye with Retisert within 36 months prior to study Day 1
* Prior intravitreal treatment of study eye with Ozurdex within 6 months prior to study Day 1
* Prior intravitreal treatment of study eye with Triesence or Trivaris within 3 months prior to study Day 1
* Prior peri-ocular or subtenon steroid treatment of study eye within 3 months prior to study Day 1
* Subjects requiring chronic systemic or inhaled corticosteroid therapy (>15mg prednisone daily) or chronic systemic immunosuppressive therapy
* Excluding certain skin cancers (specifically, basal cell carcinoma and squamous cell carcinoma), any malignancy receiving treatment, or in remission less than 5 years prior to study Day 1
* Subjects who have tested positive for human immune deficiency virus (HIV), tuberculosis or syphilis
* Systemic infection within 30 days prior to study Day 1
* Any severe acute or chronic medical or psychiatric condition that could increase the risk associated with study participation or could interfere with the interpretation of study results and, in the judgment of the investigator, could make the subject inappropriate for entry into this study
* Any other systemic or ocular condition which, in the judgment of the investigator, could make the subject inappropriate for entry into this study
* Treatment with an investigational drug or device within 30 days prior to study Day 1
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in this protocol from at least 14 days prior to study Day 1 until the Month 12 Visit
* Subjects unlikely to comply with the study protocol or who are likely to be lost to follow-up within three years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Leonin Jr., MD, Study Director — EyePoint Pharmaceuticals, Inc.
Locations (15):
- India (15):
  - LV. Prasad Eye Institute, Hyderabad, Andhra Pradesh
  - Sri Sankaradeva Nethralaya, Guwahati, Guwahati, Assam
  - Regional Institute of Opthalmology, Patna, Bihar
  - C.H. Nagri Municipal Eye Hospital, Ahmedabad, Gujarat
  - Seth G.S. Medical College & K.E.M Hospital, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital, Pune, Pune, Maharashtra
  - PBMA'S, H. V. Desai Eye Hospital, Pune, Maharashtra
  - Dr. Shroff's Charity Eye Hospital, Daryāganj, New Delhi
  - Sankara Nethralaya hospital, Chennai, Tamil Nadu
  - Vasan Eye Care Hospital, Chennai, Tamil Nadu
  - Sri Ramachandra Hospital, Chennai, Tamil Nadu
  - J L Rohatgi Memorial Eye Hospital, Kanpur, Uttar Pradesh
  - King George's Medical University, Lucknow, Uttar Pradesh
  - ICARE Eye Hospital and Research centre, Noida, Uttar Pradesh
  - Regional Institute of Ophthalmology, Kolkata, West Bengal

REFERENCES:
- [Derived] Biswas J, Tyagi M, Agarwal M; PSV-FAI-005 Investigation Group. The 0.2-mug/day Fluocinolone Acetonide Intravitreal Implant in Chronic Noninfectious Posterior Uveitis: A 3-year Randomized Trial in India. Ophthalmol Sci. 2023 Sep 16;4(1):100403. doi: 10.1016/j.xops.2023.100403. eCollection 2024 Jan-Feb. PMID 38027419

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Injection: Placebo Injection
- FAI Insert: Fluocinolone Acetonide Intravitreal (FAI) Insert Group
Period: Overall Study
Arm/Group | Sham Injection | FAI Insert
Started | 52 | 101
Completed | 24 | 67
Not Completed | 28 | 34

BASELINE CHARACTERISTICS:
Population: A total of 153 subjects were randomly assigned to 1 of 2 treatment groups: 101 subjects in the FAI insert treatment group and 52 subjects in the sham injection treatment group.
Groups:
- FAI Insert: FAI Insert Group
- Total: Total of all reporting groups
Arm/Group | Sham Injection | FAI Insert | Total
Number analyzed (Participants) | 52 | 101 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (13.74) | 39.9 (12.87) | 40.1 (13.13)
Age, Customized [Count of Participants; unit: Participants]
  <20 years | 2 | 0 | 2
  20 to <40 years | 25 | 57 | 82
  40 to <60 years | 21 | 34 | 55
  >=60 years | 4 | 10 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 62 | 96
  Male | 18 | 39 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 52 | 101 | 153
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 49 | 96 | 145
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Intention To Treat (ITT) Population [Count of Participants; unit: Participants] | 52 | 101 | 153

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence of Uveitis in Study Eye Within 6 Months
Description: Proportion of Subjects with Recurrence of Uveitis in the Study Eye within 6 Months Including Reason for Imputed Recurrence (ITT Population)
Time Frame: 6 Months
Population: Proportion of Subjects with Recurrence of Uveitis in the Study Eye within 6 Months Including Reason for Imputed Recurrence (ITT Population)
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Injection | FAI Insert
Number analyzed (Participants) | 52 | 101
Participants | 28 | 22

2. Secondary Outcome: Number of Participants With Recurrence of Uveitis in Study Eye Within 36 Months
Description: Proportion of Subjects with Recurrence of Uveitis in the Study Eye at 36 Months Including Reason for Imputed Recurrence (ITT Population)
Time Frame: 36 Months
Population: Proportion of Subjects with Recurrence of Uveitis in the Study Eye at 36 Months Including Reason for Imputed Recurrence (ITT Population)
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Injection | FAI Insert
Number analyzed (Participants) | 52 | 101
Participants | 39 | 47

ADVERSE EVENTS:
Time Frame: 36 months. All Adverse Event (AE)s will be evaluated from their onset until resolution, stabilization, last day of participation in the study of the patient or the last day of the study, whichever is first.
Description: Treatment-Emergent Ocular Adverse Events through Month 36 Visit by Eye, System Organ Class, and Preferred Term in More than 5% of Subjects in Either Treatment Group (Safety Population)
Arm/Group | Sham Injection | FAI Insert
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/101
Serious Adverse Events (participants affected / at risk) | 7/52 | 21/101
Other Adverse Events (participants affected / at risk) | 49/52 | 94/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Injection (N=52) | FAI Insert (N=101)
Cataract (Eye disorders) | 0 | 2
Choroiditis (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 2
Hypotony of eye (Eye disorders) | 0 | 8
Optic atrophy (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Uveitis (Investigations) | 1 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Vitreous haze (Eye disorders) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Tuberculosis Gastrointestinal (Infections and infestations) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Injection (N=52) | FAI Insert (N=101)
Anterior chamber cell (Eye disorders) | 7 | 10
Cataract (Eye disorders) | 10 | 17
Cataract subcapsular (Eye disorders) | 9 | 36
Conjunctival haemorrhage (Eye disorders) | 1 | 6
Cystoid macular oedema (Eye disorders) | 8 | 4
Dry eye (Eye disorders) | 2 | 5
Eye pain (Eye disorders) | 8 | 6
Eye pruritus (Eye disorders) | 6 | 4
Glaucoma (Eye disorders) | 1 | 5
Hypotony of eye (Eye disorders) | 0 | 10
Iris adhesions (Eye disorders) | 4 | 2
Macular fibrosis (Eye disorders) | 0 | 7
Macular oedema (Eye disorders) | 11 | 9
Ocular hyperaemia (Eye disorders) | 4 | 2
Posterior capsule opacification (Eye disorders) | 5 | 9
Uveitis (Eye disorders) | 27 | 20
Visual acuity reduced (Eye disorders) | 4 | 15
Vitreous haze (Eye disorders) | 9 | 12
Vitritis (Eye disorders) | 10 | 9
Intraocular pressure increased (Investigations) | 2 | 32
Conjunctivitis (Infections and infestations) | 4 | 4
Furuncle (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Tuberculosis gastrointestinal (Infections and infestations) | 1 | 0
Typhoid fever (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Asthenia (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Hypertension (Vascular disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Parkinsonism (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperprolactinaemia (Endocrine disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Breast discharge (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT02746991/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT02746991/SAP_002.pdf